CLINICAL TRIAL: NCT05774899
Title: A Phase 1/2 Study of CB-103 (Oral Pan-NOTCH Inhibitor) With Abemaciclib or Lenvatinib in Combination in Patients With NOTCH Activated Adenoid Cystic Carcinoma (CALCulus)
Brief Title: CB-103 With Either Lenvatinib or Abemaciclib in Patients With NOTCH ACC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Glenn J. Hanna (Other)
Collaborators: Adenoid Cystic Carcinoma Research Foundation (Other); Cellestia Biotech AG (Industry)
Responsible Party: Sponsor-Investigator, Glenn J. Hanna, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-011
Record Dates: First submitted 2023-03-14; First posted 2023-03-20 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Adenoid Cystic Carcinoma; Metastatic Adenoid Cystic Carcinoma; Recurrent Adenoid Cystic Carcinoma
Keywords: Adenoid Cystic Carcinoma; Metastatic Adenoid Cystic Carcinoma; Recurrent Adenoid Cystic Carcinoma; ACC
MeSH Terms: conditions — Carcinoma, Adenoid Cystic | interventions — abemaciclib; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Experimental: Cohort 1A - CB-103 + Abemaciclib (Experimental): A modified 3+3 dose escalation design will be used. 3-9 participants will receive:
  * Standard of care Abemaciclib.
  * Cycle 1 - End of Treatment
    --Days 1- 28 of 28-day cycle: Predetermined dose of CB-103 2x daily on five consecutive days followed by two days of treatment break in each treatment week.
  * A safety review will be performed by primary investigation after completion of the ramp-up phase.
  Interventions: Drug: CB-103; Drug: Abemaciclib
- Experimental: Cohort 1B - CB-103 + Abemaciclib (Experimental): Participants will receive:
  * Cycle 1 - End of Treatment
    --Days 1- 28 of 28-day cycle: Predetermined dose of CB-103 2x daily on five consecutive days followed by two days of treatment break in each treatment week and predetermined dose of Abemaciclib 1x daily.
  * Therapy will continue until disease progression, therapy intolerance, or participant withdrawal.
  * End of Treatment (EOT) visit within 30 days of last administration of study treatments.
  Interventions: Drug: CB-103; Drug: Abemaciclib
- Experimental: Cohort 2A- Lenvatinib + CB-103 (Experimental): A modified 3+3 dose escalation design will be used. 3-9 participants will receive:
  * Standard of care VEGFR TKI.
  * Cycle 1 - End of Treatment
    --Days 1- 28 of 28-day cycle: Predetermined dose of CB-103 2x daily on five consecutive days followed by two days of treatment break in each treatment week.
  * A safety review will be performed by primary investigation after completion of the ramp-up phase.
  Interventions: Drug: CB-103; Drug: Lenvatinib
- Experimental: Cohort 2B- Lenvatinib + CB-103 (Experimental): Participants will receive:
  * Continue standard of care VEGFR TKI at prior dose and schedule.
  * Cycle 1 - End of Treatment
    --Day 1- 28 of 28-day cycle: Predetermined dose of CB-103 2x daily on five consecutive days followed by two days of treatment break in each treatment week.
  * Therapy will continue until disease progression, therapy intolerance, or participant withdrawal.
  * End of Treatment (EOT) visit within 30 days of last administration of study treatments.
  Interventions: Drug: CB-103; Drug: Lenvatinib

INTERVENTIONS:
Drug: CB-103 — First-in-class pan-NOTCH inhibitor, capsule taken orally.
Drug: Abemaciclib — CDK4/6 inhibitor, tablet taken orally.
  Arms: Experimental: Cohort 1A - CB-103 + Abemaciclib; Experimental: Cohort 1B - CB-103 + Abemaciclib
Drug: Lenvatinib — Per standard care, capsule taken orally.
  Other Names: Lenvima
  Arms: Experimental: Cohort 2A- Lenvatinib + CB-103; Experimental: Cohort 2B- Lenvatinib + CB-103

SUMMARY:
The goal of this study is to treat patients with NOTCH active advanced adenoid cystic carcinoma (ACC) tumors with a combination or two different oral medications to slow tumor growth and improve survival outcomes.

The names of the study drugs involved in this study are:

* CB-103 (an oral NOTCH pathway inhibitor)
* Abemaciclib (CDK4/6 inhibitor)
* Lenvatinib (a vascular endothelial growth factor receptor (VEGFR) tyrosine kinase inhibitor (TKI))

DETAILED DESCRIPTION:
This is a phase 2, open-label, non-randomized, parallel cohort, multicenter study investigating the novel pan-NOTCH inhibitor, CB-103, in combination with the CDK4/6 inhibitor, Abemaciclib, and CB-103 in combination with the multi-targeted vascular endothelial growth factor receptor (VEGFR) tyrosine kinase inhibitor (TKI), Lenvatinib for patients with advanced, incurable, or metastatic adenoid cystic carcinoma (ACC) with a Notch pathway activating mutation.

Participants will be placed into one of two treatment groups: Cohort 1: CB-103 + Abemaciclib or Cohort 2: VEGFR TKI Lenvatinib + CB-103.

The U.S. Food and Drug Administration (FDA) has not approved CB-103 as a treatment for any disease.

The FDA has not approved Abemaciclib or Lenvatinib for advanced adenoid cystic carcinoma (ACC)), but it has been approved for other uses or cancer types.

Study procedures include screening for eligibility, treatment visits, radiologic scans of tumors, and blood tests.

Participation in this study is expected to last about 2 years or until disease progression, therapy intolerance, or participant withdrawal.

It is expected that about 32 people will take part in this research study.

Cellestia Biotech AG is supporting this research study by providing funding.

ELIGIBILITY:
Participants must meet the following eligibility criteria at the time of screening to be eligible to participate in the study:

Eligibility Criteria

1. Participants must have histologically confirmed adenoid cystic carcinoma (ACC) with evidence of recurrent, metastatic or advanced, incurable disease arising from any primary site
2. Activating mutation in the NOTCH signaling pathway
3. In Cohort 1 only, prior multitargeted VEGFR TKI or systemic therapy is permitted.
4. In Cohort 2 only, no prior multitargeted VEGFR TKI therapy is permitted, but prior systemic chemotherapy as part of definitive or curative intent management is permitted.

   a. Any participant must obtain prior approval from insurance to reimburse for oral Lenvatinib, or off-label drug assistance to secure Lenvatinib for the duration of the study or agree to self-pay for oral Lenvatinib or obtain institutional commitment from the study site to provide Lenvatinib.
5. Age 18 years or older
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
7. Patients able and willing to swallow oral capsules or tablet medications.
8. At least one measurable lesion (RECIST v1.1)
9. Participant must have organ and marrow function as defined below within 14 days prior to study registration (ULN=upper limit of normal per institution):

   Absolute neutrophil count (ANC) ≥1.5 x 109/L Hemoglobin (Hgb) ≥9 g/dL (patients may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after the erythrocyte transfusion).

   Platelet count ≥100 x 109/L (without transfusion within the last 5 days) Serum creatinine ≤1.5x ULN or serum creatinine clearance (CrCl) ≥50 mL/min (estimated by Cockcroft-Gault formula) Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3x ULN Total serum bilirubin ≤1.5x ULN (patients with Gilbert's syndrome with a total bilirubin ≤2.0 times ULN and direct bilirubin within normal limits are permitted).
10. Baseline proteinuria with a urinalysis or urine dipstick value of 2+ requires a spot urine protein/creatinine ratio of <0.3 (or 24-hour urine collection protein value <300 mg/g) in Cohort 2 only
11. Participants with treated brain or CNS metastases are eligible if follow-up brain imaging after CNS-directed therapy shows no convincing evidence of progression and patients are neurologically stable with no new neurological deficits.
12. Female subjects of childbearing potential should have a negative serum pregnancy test within 7 days before start of study treatment.
13. Female and male subjects of childbearing potential must agree to use an adequate method of contraception to avoid pregnancy (with at least 99% certainty) from screening through 90-days or 3-months post-treatment completion (see Appendix B).
14. Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
15. Patients who received chemotherapy must have recovered (CTCAE grade ≤1) from the acute effects of chemotherapy except for residual alopecia or grade 2 peripheral neuropathy. A washout period of at least 21 days is required between last chemotherapy dose and start of therapy (provided the patient did not receive radiotherapy).

Exclusion Criteria

1. Participant has untreated or clinically symptomatic CNS metastases and/or carcinomatous meningitis
2. The patient has had major surgery within 14 days prior to study registration.
3. The patient has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment, history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline grade 2 or higher diarrhea).
4. Impairment of GI function or presence of GI disease that may significantly alter the absorption of the study agents (e.g. ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
5. The patient has active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Screening is not required for enrollment.
6. The patient has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest
7. Pregnant or lactating women. Pregnant women are excluded from this study because of the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued.
8. Patients who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and start of therapy. Patients on anticoagulants that require INR monitoring (such as warfarin). The patient has received an experimental treatment in a clinical trial within the last 30 days or 5 half-lives, whichever is longer, or is currently enrolled in any other type of medical research judged by the sponsor not to be scientifically or medically compatible with this study.
9. Corrected QTcF >450 msec for males and >470 msec for females in screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) of Cohort 1 | At 4 months
  Progression-Free Survival (PFS) is defined as the time from study registration to the earlier of progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation. Median PFS will be estimated via the Kaplan-Meier method to estimate all time-to-event endpoints with corresponding 95% confidence intervals (CI) for the median or time-specific event time
Progression-Free Survival (PFS) of Cohort 2 | At 4 months
  Progression-Free Survival (PFS) is defined as the time from study registration to the earlier of progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation.

SECONDARY OUTCOMES:
Number of Participants with treatment related Adverse Events per CTCAE 5.0 | Up to 2 years
  Assessed using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Overall Response Rate (ORR) | From enrollment to end of treatment up to 2 years
  Per RECIST v1.1
Overall Survival (OS) | Up to 2 years
  Overall Survival (OS) is defined as the time from study registration to death due to any cause, or censored at date last known alive.
Duration of Overall Response (DOR) | Up to 2 years
  The duration of overall response is measured from the time measurement criteria are met for Complete Response (CR) or Partial Response (PR), whichever is first recorded, until the first date that recurrent or progressive disease is objectively documented. Participants without events reported are censored at the last disease evaluation).

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Hanna, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu